CLINICAL TRIAL: NCT05403736
Title: IIT2021-07-Atkins-CARMA: Cardiac Aggressive Risk Mitigation in Thoracic Radiotherapy (CARMA) Trial
Brief Title: Cardiac Aggressive Risk Mitigation in Thoracic Radiotherapy (CARMA) Trial
Acronym: CARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Katelyn Atkins, Assistant Professor, Radiation Oncology, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2021-07-Atkins-CARMA
Record Dates: First submitted 2022-03-11; First posted 2022-06-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: radiation therapy; cardio-oncology; cardiology; cardiac toxicity; lung cancer; esophageal cancer; breast cancer; thoracic radiotherapy
MeSH Terms: conditions — Neoplasms; Cardiotoxicity; Lung Neoplasms; Esophageal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CARMA (Experimental): Cardiac Aggressive Risk MitigAtion plan with biosensor monitoring
  Interventions: Other: Cardiac Aggressive Risk MitigAtion Plan

INTERVENTIONS:
Other: Cardiac Aggressive Risk MitigAtion Plan — Cardio-oncology consultation along with long-term collaborative cancer care visits during standard of care radiation therapy that will occur weekly for up to 6 weeks followed by 6-week and 3-month follow-up visits. Health will be monitored with biosensor monitoring devices.
  Other Names: FitBit; Omron EVOLV Automatic Blood Pressure Monitor; AliveCor KardiaMobile Personal EKG Monitor; cardio-oncology consultation

SUMMARY:
The purpose of this study is to examine adherence to cardio-oncology consultation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate patient participation in a plan to improve heart health after radiation therapy by having a cardio-oncology assessment early during cancer treatment. Cardiologists and cancer doctors will review any cardiovascular risk factors (heart conditions, hypertension, bleeding disorders, smoking history, obesity, cholesterol and diabetes) and develop a personalized treatment plan. In addition, the study will evaluate use of wearable devices such as a FitBit, and remote EKG (Omron EVOLV) and blood pressure monitoring (AliveCor KardiaMobile) devices to monitor participant's health. Blood will be drawn at three separate timepoints for biomarker testing of heart injury, aging, inflammation and metabolism.

Study visits will occur at baseline, weekly during radiation therapy, 6 weeks and 3 months after completion of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any stage (I-IV) malignancy being treated with high dose (≥30 Gy) radiotherapy where the heart is in the treatment field.
* Have Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
* Planning to receive standard of care radiotherapy treatments.
* Access to a smart device that has the capability to sync to the devices.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Ability to read, write and understand English.

Exclusion Criteria:

* Known allergy to surgical steel or elastomer/rubber.
* Heart attack within 6 months prior to study enrollment.
* Severe and/or active scleroderma or systemic lupus erythematosus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete the cardio-oncology consultation visit | From baseline to 3 months
  Adherence is defined as 70% of the participants completing the cardio-oncology consultation visit prior to or during radiotherapy.

SECONDARY OUTCOMES:
Number of participants who wear the FitBit device at least 10 hours per day for 4 out of the 7 days prior to each study visit | From baseline to 3 months
  Proportion of participants who wear the FitBit device at least 10 hours per day for 4 out of the 7 days prior to each study visit
Number of participants who obtain blood pressure readings for at least 4 timepoints | From baseline to 3 months
  Proportion of participants who obtain blood pressure readings for at least 4 timepoints.
  -The Omron blood pressure monitor will be used to obtain blood pressure readings.
Number of participants who obtain electrocardiogram (EKG) readings for at least 4 timepoints | From baseline to 3 months
  Proportion of participants who obtain EKG readings for at least 4 timepoints.
  -The AliveCor KardiaMobile EKG monitor will be used to obtain EKG readings
Rate of cardiovascular therapeutic medication intervention recommendations by the cardio-oncologist | From baseline to 3 months
  Number of participants provided recommendation to either initiate, or modify the dose of, a cardiovascular risk-reducing medication (anti-lipid, anti-platelet, anti-coagulation, anti-hypertensive). Expressed as the number of participants as a fraction of the total number of participants.
Rate of compliance with cardiovascular therapeutic medication intervention | From baseline to 3 months
  Compliance will be assessed by self-reporting of medication usage at the 3-month follow-up and defined as yes or no for all recommended cardiovascular therapeutic medication interventions. Expressed as the number of participants as a fraction of the total number of participants.
Evaluate participant intervention perspectives at the end of the study. | At 3 months
  * Analyze participate attitudes and perspectives on implementation and impact of the cardiovascular intervention plan. Participants will be asked to complete a survey at the 3-month visit.
  * Each question is either answered on a scale of 1-4 or strongly agree-strongly disagree, where higher scores indicate the highest level of burden or disagreement, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Atkins, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cancer Clinical Trials Office, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data (including data dictionaries) supporting the manuscript findings will be shared beginning three months after publication and without end date with qualified investigators whose proposed use of the data has been approved by an institutional review board and following execution of a data use agreement per Cedars-Sinai Medical Center institutional policy. The study protocol will additionally be shared.